CLINICAL TRIAL: NCT03998982
Title: A Single-center Prospective Randomized Study of Glycyrrhetinic Acid Combined With Dexamethasone in the Treatment of Newly Diagnosed Primary Immune Thrombocytopenia (ITP)
Brief Title: Glycyrrhetinic Acid Combined With Dexamethasone in Management of Newly Diagnosed ITP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Glycyrrhetinic Acid+DXM in ITP
Record Dates: First submitted 2019-06-25; First posted 2019-06-26 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Immune Thrombocytopenia
Keywords: ITP；glycyrrhetinic acid；dexamethasone
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Glycyrrhetinic Acid; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- glycyrrhetinic acid Combining HD-DXM (Active Comparator): Compound glycyrrhizin tablets 75mg three times per day, 1 month, and HD-DXM (orally at 40 mg daily for 4d )
  Interventions: Drug: Glycyrrhetinic Acid; Drug: Dexamethasone
- HD-DXM (Active Comparator): HD-DXM (orally at 40 mg daily for 4d )
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Glycyrrhetinic Acid — Compound glycyrrhizin tablets 75 mg three times per day, 1 month
  Arms: glycyrrhetinic acid Combining HD-DXM
Drug: Dexamethasone — HD-DXM (orally at 40 mg daily for 4d)

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University in China. In order to report the efficacy and safety of glycyrrhetinic acid combining with high-dose dexamethasone for the treatment of adults with newly-diagnosed primary immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators anticipate to undertaking a parallel group, single-centre, randomised controlled trial of 30 ITP adult patients. One part of the participants are randomly selected to receive glycyrrhetinic acid (given compound glycyrrhizin tablets orally at a dose of 225mg per day for 1 month), combining with dexamethasone (given orally at a dose of 40 mg per day for 4 days, two-cycles with an interval of 10 days); the others are selected to receive high-dose of dexamethasone treatment plus placebo. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study. In order to report the efficacy and safety of glycyrrhetinic acid combining with high-dose dexamethasone therapy for the treatment of adults with ITP.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for immune thrombocytopenia;
* Untreated hospitalized patients, may be male or female, between the ages of 18~ 80 years;
* To show a platelet count <30 * 10^9/L, and with bleeding manifestations;
* Willing and able to sign written informed consent

Exclusion Criteria:

* Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit;
* Received second-line ITP-specific treatments (eg, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) within 3 months before the screening visit;
* Received high-dose steroids or IVIG in the 3 weeks prior to the start of the study;
* Current HIV infection;
* Severe medical condition (lung, hepatic or renal disorder) other than chronic ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac
* Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period;
* Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test;
* Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2021-06-10 (Estimated); Study Completion 2021-06-10 (Estimated)

PRIMARY OUTCOMES:
Sustained response to ITP treatments | 3 months after treatment started
  Percentage of patients maintaining PLT count over 30*10^9 without bleeding

SECONDARY OUTCOMES:
Evaluation of platelet response | 3 months after treatment started
  Complete response (CR)# A platelet count ≥ 100 * 10^9/L measured on two occasions > 7 days apart and the absence of bleeding. Response (R)# A platelet count ≥ 30 * 10^9/L and a greater than two fold increase in platelet count from baseline measured on two occasions > 7 days apart and the absence of bleeding. No response (NR)# A platelet count < 30 * 10^9/L or a less than two fold increase in platelet count from baseline or the presence of bleeding. Platelet count must be measured on two occasions more than a day apart.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, MD,PhD, Principal Investigator — Shandong University Qilu Hospital
Locations (1):
- Qilu hospital, Shandong University, Jinan, Shandong, China